CLINICAL TRIAL: NCT02658513
Title: Evaluation of Lancet Blood Sampling for Radioiodine Dosimetry in Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, James Scuffham, Clinical Scientist, Royal Surrey County Hospital NHS Foundation Trust
Other Study IDs: 14OncN0013
Record Dates: First submitted 2015-12-24; First posted 2016-01-20 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Cancer of the Thyroid; Cancer of Thyroid; Thyroid Cancer; Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Patients: All patients will undergo both of the following interventions:
  Lancet blood sampling Standard intravenous blood sampling
  Interventions: Other: Lancet blood sampling; Other: Standard intravenous blood sampling

INTERVENTIONS:
Other: Lancet blood sampling — Blood samples will be obtained using a finger-prick (lancet) technique.
Other: Standard intravenous blood sampling — Blood samples will be obtained using a standard intravenous technique.

SUMMARY:
Recently published European guidance recommends the evaluation of the radiation dose to the bone marrow in patients undergoing radioiodine therapy for thyroid cancer. The methods described in these guidelines require serial blood samples to be taken from the patient, followed by a sophisticated analysis to determine the radiation dose. However, radiation risk assessments carried out locally have indicated that a relatively high radiation exposure will be received by the operator taking the blood samples, which may prohibit this procedure being carried out routinely.

The radiation dose to the operator will be lowered if the duration of the blood sampling procedure were reduced. The investigators hypothesize that the use of a lancet and pipette to collect blood from the finger tip will greatly reduce the time spent in proximity to the patient, significantly reducing the operator exposure and allowing this procedure to be performed routinely. The proposed method is also less invasive for the patient compared to the intravenous sampling recommended in the guidelines. A proof-of-principal pilot project using radioiodine diluted to the expected concentration in blood has indicated that using very small volumes of blood (such as from a lancet) does not compromise the accuracy of the dosimetry measurement when compared to large-volume standard blood samples.

The primary aim of this study is to investigate whether sampling a small volume of blood using a lancet and pipette can replace standard intravenous blood samples for bone marrow dosimetry in patients undergoing radioiodine treatment for thyroid cancer. Statistical tests will determine whether there is a significant difference between the doses calculated using each blood sampling method. In addition, the investigators will measure the radiation exposure received by the operator during each procedure using Electronic Portable Dosimeters. The results of these measurements will be used to quantify the reduction in operator radiation exposure afforded by the new technique.

DETAILED DESCRIPTION:
Recruitment:

Patients will be recruited to the trial from the pool of routine referrals for this therapy. Potential participants will receive an information leaflet via the post several weeks in advance of attendance at clinic. Patients will have the opportunity to telephone the study team during this time to answer any questions. Patients who are interested in participating will have the procedure further explained verbally by a physicist on the study team upon attending for therapy. The patient will then have time to consider whether or not to participate in the study. Written consent will be sought before commencing the therapy.

Procedures:

In light of the recent guidelines, the proposed new clinical protocol will include blood samples taken from the patient during the in-patient stay. On the day of treatment, blood samples will be taken at 2h and 6h after radioiodine administration, at the same time as the clearance measurements. Thereafter, a blood sample will be taken from the patient once per day, at the same time as one of the clearance measurements. In addition, a further blood sample will be taken when the patient attends for whole-body and SPECT/CT scans. These blood samples will then be analysed in the laboratory using standard radiation measurement procedures to determine the blood dose according to the European guidelines.

This study will involve the patient having blood samples taken by two different methods at each of the time points described above. In the first method, a butterfly needle will be used to gain intravenous access at the antecubital fossa, and a heparinised vacutainer will be used to collect a 4ml blood sample. The needle will then be removed and the venepuncture site dressed with a plaster. In the second method, a single-use safety lancet will be used to puncture the skin on the finger, and a small pipette used to collect a small quantity of blood. The entire pipette will be transferred to a sample tube for later processing. The puncture site on the finger will then be dressed with a small plaster. The exact start and end times for each sample will be recorded using a radio-controlled standard clock.

While carrying out blood sampling, the operator will wear an electronic portable dosimeter (EPD) to measure radiation exposure. This device will be positioned on the operator's chest to reflect the whole body dose received, and will be configured to record the radiation dose as a function of time during the procedure. After the procedure, the data from the EPD will be downloaded and split into two segments representing each blood sampling procedure, using the recorded timing information. Each segment will then be integrated to give the total radiation exposure received by the operator for each procedure. At the end of the treatment, patients will be asked which of the two blood sampling methods were the most tolerable.

Each sample will be labelled with the patient identification number, the date, time and radioisotope (I-131). To minimise the risk of spills, the samples will be transferred to a tray and moved to the Nuclear Medicine Department using a trolley. Sample manipulations will be carried out in the low level counting laboratory in the Nuclear Medicine Department. Three 1ml aliquots of whole blood will be removed from each vacutainer and transferred to appropriately labelled sample containers using an Eppendorf pipette. The volume of the samples collected by pipette will be determined by measuring the weight of the sample and subtracting the previously determined combined weight of the empty pipette and sample tube. Once all the blood samples have been collected and processed, measurements will be taken in an automated gamma counter to determine the concentration of radioiodine. The counting time for the pipette samples will be increased compared to the intravenous samples, in order to ensure the final dosimetry calculations are not influenced by the statistical uncertainty in the measured counts from the smaller volume samples. The resulting data will then be used in the detailed dosimetry calculations, in accordance with the published European guidelines.

Sample Size:

There is no published data available on the intra-patient variation of bone marrow dose using either of the two proposed blood sampling methods. Without knowledge of the expected variances of the measurements in question, accurate sample size calculations are not possible prior to commencing the study. A sample size of 35 patients will be used in this pilot study - this sample size was chosen based on the number of patients seen in the department for this therapy. Recruiting a sample size of 35 patients is achievable within a 2 year time frame. However, the study will be stopped early if the total annual radiation exposure to the operators, combined with the total radiation exposure due to normal clinical workload, is likely to exceed the annual UK dose constraint of 2mSv for whole body radiation exposure (The Ionising Radiations Regulations 1999, SI 1999/3232).

Data Analysis:

Using the measured concentrations of radioiodine in the blood samples, the radiation dose to the bone marrow of each participant will be calculated following the methods described in European guidance (Luster et al, Eur J Nucl Med Mol Imaging 35(10) 1941 2008). This calculation will be performed for each of the two blood sampling methods, creating paired measurements of the same variable for each participant. The statistical significance of the percentage difference in bone marrow dose calculated from each blood sampling method will then be assessed using a Wilcoxon matched pairs test with the null hypothesis that there is no difference in the calculated bone marrow doses. This study has 80% power to demonstrate at the 5% level of statistical significance a difference of no less than 5% between the mean values for the two bone marrow doses. Therefore statistical analysis of the differences has 80% power to show that the null hypothesis that the difference is no greater than 5% is tenable, if indeed this null hypothesis holds true in the population.

The radiation exposure received by the operator during each blood sampling procedure will be measured using an Electronic Portable Dosimeter (EPD) worn on the chest of the operator. The data will be split into two using the known start and end times of each blood sampling procedure. The data will then be integrated over each time period to calculate the total radiation dose for each interval. This will create paired measurements of the same variable for each blood sampling event for each participant. The statistical significance of the percentage difference in the radiation exposures received by the operator during each blood sampling method will then be assessed using a Wilcoxon matched paired test with the null hypothesis that there is no difference between the measured radiation doses. The aim in this case is to show statistically that the null hypothesis of no difference in the mean radiation doses for the 2 techniques is untenable.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing inpatient radioiodine therapy for thyroid cancer

Exclusion Criteria:

* Pregnant or breastfeeding women
* Paediatric patients
* Patients with known trypanophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid cancer receiving radioiodine therapy after total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Quantify the bone marrow doses (in Gray) for each of the two blood sampling techniques. | Within 1 month of completing recruitment

SECONDARY OUTCOMES:
Quantify the radiation exposure (in milli-Sieverts) to staff for each of the two blood sampling techniques. | Within 1 month of completing recruitment

CONTACTS AND LOCATIONS:
Overall Officials: James W Scuffham, PhD, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (1):
- Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No